CLINICAL TRIAL: NCT00900224
Title: Assessment of Novel Molecular Markers in Acute Myeloid Leukemia
Brief Title: Studying Tissue and Blood Samples From Patients With Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-20202; CALGB-20202; CDR0000617738 (Registry Identifier: NCI Physician Reference Desk)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — DNA Methylation; Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Chromatography, High Pressure Liquid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow aspirate, whole blood, buccal cell sample and bone marrow biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Previously procured and archived bone marrow aspirate samples, blood and buccal cell samples, and bone marrow biopsy slides are analyzed for FLT3 ITD, MLL PTD, NPM1, KIT, KRAS, NRAS, CEBPA, WT1, JAK2, RUNX1, TET2, ASXL1, IDH1 and IDH2, CBL, and DNMT3A mutations, CBF fusion genes, levels of BAALC, ERG, EVI1, MN1, and APP microarray gene-expression, microRNA gene-expression signature, levels of methylation of genes silenced in AML, and genomic DNA by PCR amplification, RT-PCR, and denaturing high-performance liquid chromatography.
  Interventions: Genetic: DNA analysis; Genetic: DNA methylation analysis; Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: polymerase chain reaction; Genetic: reverse transcriptase-polymerase chain reaction; Other: high performance liquid chromatography; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: high performance liquid chromatography
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tissue and blood samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Prospectively obtain specimens required for diagnostic review and molecular characterization ensuring eligibility for CALGB Leukemia Committee Clinical trials (for clinical trials designed to enroll specific molecular subtypes, results to determine eligibility will be reported to treating physicians no more than 72 hours after specimen receipt at the repository).
* Determine the frequency of specific gene markers (i.e., FLT3 ITD, CBF, MLL PTD, NPM1, KIT, RAS, CEBPA, WT1, JAK2, RUNX1, TET2, CBL, IDH1 and IDH2, ASXL1, mutations, aberrant BAALC, ERG, FLT3, MN1, EVI1, and APP) over-expression and levels of promoter methylation of specific genes (e.g., ESR1, WIT1, P15, MYOD1, ID4, DPK) in defined cytogenetic subgroups of patients with acute myeloid leukemia (AML).
* Correlate these gene markers with clinical and laboratory parameters in these patients.
* Correlate these gene markers with clinical outcome (i.e., complete remission [CR], disease-free survival [DFS], cumulative incidence of relapse [CIR], and overall survival [OS]) in these patients.
* Identify specific microarray multi-gene expression signatures in these patients.
* Correlate specific microarray multi-gene expression signatures with clinical and laboratory parameters in these patients.
* Correlate specific microarray multi-gene expression signatures with clinical outcome (i.e., CR, DFS, CIR, and OS) in these patients.
* Identify specific microarray multi-microRNA (miR) expression signatures in these patients
* Correlate specific microarray multi-miR expression signatures with clinical and laboratory parameters in these patients.
* Correlate specific microarray multi-miR expression signatures with clinical outcome (i.e., CR, DFS, CIR, and OS) in these patients.
* Explore the relative contribution of prognostic gene markers (i.e., FLT3 ITD, MLL PTD, NPM1, KIT, RAS, CEBPA, WT1, and JAK2 mutations, and aberrant BAALC, ERG, FLT3, MN1, and EVI1 over-expression), levels of promoter methylation of specific genes (e.g., ESR1, WIT1, P15, MYOD1, ID4, DPK), and microarray gene and miR expression signatures in defined cytogenetic subgroups of AML.
* Determine changes in these molecular markers and microarray gene and miR expression signatures at CR and relapse and the influence that these changes have on subsequent clinical course.
* Correlate the relative level of nuclear pSTAT5 and pERK in bone marrow blasts with outcome (EFS, CR, DFS, OS).

OUTLINE: This is a multicenter study.

Previously procured and archived bone marrow aspirate samples, blood and buccal cell samples, and bone marrow biopsy slides are analyzed for FLT3 ITD, MLL PTD, NPM1, KIT, KRAS, NRAS, CEBPA, WT1, JAK2, RUNX1, TET2, ASXL1, IDH1 and IDH2, and CBL mutations, CBF fusion genes, levels of BAALC, ERG, EVI1, MN1, and APP microarray gene-expression, microRNA gene-expression signature, levels of methylation of genes silenced in AML, and genomic DNA by PCR amplification, RT-PCR, and denaturing high-performance liquid chromatography.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (AML)
* Tissue samples from previously untreated patients with AML considered for enrollment onto ongoing and future CALGB treatment protocols
* AML tissue samples from companion Leukemia Tissue Bank protocol CALGB-9665 and the companion cytogenetic protocol CALGB-8461
* AML diagnostic bone marrow and/or blood samples from patients enrolled on CLB-9720, CLB-9621 (all cytogenetic subtypes), and CALGB-19808 (abnormal cytogenetics only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Presence of molecular markers that fulfill eligibility criteria in diagnostic samples from AML patients considered for CALGB therapeutic protocols | baseline
Frequency of specific single-gene markers over-expression and levels of promoter methylation of specific genes | baseline
Predictive value of specific single-gene markers | baseline
Microarray multi-gene and multi-miR expression signatures | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clara Bloomfield, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (77):
- United States (77):
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Becker H, Marcucci G, Maharry K, Radmacher MD, Mrozek K, Margeson D, Whitman SP, Paschka P, Holland KB, Schwind S, Wu YZ, Powell BL, Carter TH, Kolitz JE, Wetzler M, Carroll AJ, Baer MR, Moore JO, Caligiuri MA, Larson RA, Bloomfield CD. Mutations of the Wilms tumor 1 gene (WT1) in older patients with primary cytogenetically normal acute myeloid leukemia: a Cancer and Leukemia Group B study. Blood. 2010 Aug 5;116(5):788-92. doi: 10.1182/blood-2010-01-262543. Epub 2010 May 4. PMID 20442368
- [Derived] Archer KJ, Fu H, Mrozek K, Nicolet D, Mims AS, Uy GL, Stock W, Byrd JC, Hiddemann W, Braess J, Spiekermann K, Metzeler KH, Herold T, Eisfeld AK. Identifying long-term survivors and those at higher or lower risk of relapse among patients with cytogenetically normal acute myeloid leukemia using a high-dimensional mixture cure model. J Hematol Oncol. 2024 May 3;17(1):28. doi: 10.1186/s13045-024-01553-6. PMID 38702786
- [Derived] Ozga M, Nicolet D, Mrozek K, Yilmaz AS, Kohlschmidt J, Larkin KT, Blachly JS, Oakes CC, Buss J, Walker CJ, Orwick S, Jurinovic V, Rothenberg-Thurley M, Dufour A, Schneider S, Sauerland MC, Gorlich D, Krug U, Berdel WE, Woermann BJ, Hiddemann W, Braess J, Subklewe M, Spiekermann K, Carroll AJ, Blum WG, Powell BL, Kolitz JE, Moore JO, Mayer RJ, Larson RA, Uy GL, Stock W, Metzeler KH, Grimes HL, Byrd JC, Salomonis N, Herold T, Mims AS, Eisfeld AK. Sex-associated differences in frequencies and prognostic impact of recurrent genetic alterations in adult acute myeloid leukemia (Alliance, AMLCG). Leukemia. 2024 Jan;38(1):45-57. doi: 10.1038/s41375-023-02068-8. Epub 2023 Nov 28. PMID 38017103
- [Derived] Rebechi M, Kohlschmidt J, Mrozek K, Nicolet D, Mims AS, Blachly JS, Orwick S, Larkin KT, Oakes CC, Hantel A, Carroll AJ, Blum WG, Powell BL, Uy GL, Stone RM, Larson RA, Byrd JC, Paskett ED, Plascak JJ, Eisfeld AK. Association of social deprivation with survival in younger adult patients with AML: an Alliance study. Blood Adv. 2023 Aug 8;7(15):4019-4023. doi: 10.1182/bloodadvances.2022009325. No abstract available. PMID 37196637
- [Derived] Mrozek K, Kohlschmidt J, Blachly JS, Nicolet D, Carroll AJ, Archer KJ, Mims AS, Larkin KT, Orwick S, Oakes CC, Kolitz JE, Powell BL, Blum WG, Marcucci G, Baer MR, Uy GL, Stock W, Byrd JC, Eisfeld AK. Outcome prediction by the 2022 European LeukemiaNet genetic-risk classification for adults with acute myeloid leukemia: an Alliance study. Leukemia. 2023 Apr;37(4):788-798. doi: 10.1038/s41375-023-01846-8. Epub 2023 Feb 23. PMID 36823396
- [Derived] Fobare S, Kohlschmidt J, Ozer HG, Mrozek K, Nicolet D, Mims AS, Garzon R, Blachly JS, Orwick S, Carroll AJ, Stone RM, Wang ES, Kolitz JE, Powell BL, Oakes CC, Eisfeld AK, Hertlein E, Byrd JC. Molecular, clinical, and prognostic implications of PTPN11 mutations in acute myeloid leukemia. Blood Adv. 2022 Mar 8;6(5):1371-1380. doi: 10.1182/bloodadvances.2021006242. PMID 34847232
- [Derived] Mims AS, Kohlschmidt J, Borate U, Blachly JS, Orwick S, Eisfeld AK, Papaioannou D, Nicolet D, Mromicronzek K, Stein E, Bhatnagar B, Stone RM, Kolitz JE, Wang ES, Powell BL, Burd A, Levine RL, Druker BJ, Bloomfield CD, Byrd JC. A precision medicine classification for treatment of acute myeloid leukemia in older patients. J Hematol Oncol. 2021 Jun 23;14(1):96. doi: 10.1186/s13045-021-01110-5. PMID 34162404
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516